CLINICAL TRIAL: NCT03912415
Title: An International Randomized Double-blind Clinical Trial of BCD-100 Plus Platinum-based Chemotherapy With and Without Bevacizumab Versus Placebo Plus Platinum-based Chemotherapy With and Without Bevacizumab as First-Line Treatment of Subjects With Advanced Cervical Cancer
Brief Title: Efficacy and Safety of BCD-100 (Anti-PD-1) in Combination With Platinum-Based Chemotherapy With and Without Bevacizumab as First-Line Treatment of Subjects With Advanced Cervical Cancer (FERMATA)
Acronym: FERMATA
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Biocad (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BCD-100-5
Record Dates: First submitted 2019-04-10; First posted 2019-04-11 (Actual); Last update posted 2020-09-18 (Actual); Status verified 2020-09

CONDITIONS: Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Bevacizumab; Paclitaxel; Cisplatin; Carboplatin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BCD-100 (Experimental): BCD-100 3 mg/kg Q3W
  Interventions: Biological: BCD-100; Biological: Bevacizumab; Drug: Paclitaxel; Drug: Cisplatin (or Carboplatin)
- Placebo (Placebo Comparator)
  Interventions: Biological: Bevacizumab; Drug: Paclitaxel; Drug: Cisplatin (or Carboplatin); Other: Placebo

INTERVENTIONS:
Biological: BCD-100 — Anti-PD-1 monoclonal antibody, IV infusion
  Arms: BCD-100
Biological: Bevacizumab — IV infusion
Drug: Paclitaxel — IV infusion
Drug: Cisplatin (or Carboplatin) — IV infusion
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This is a randomized, multicenter, double-blind, Phase 3 study of efficacy and safety of BCD-100 plus platinum-based chemotherapy with and without bevacizumab versus placebo plus platinum-based chemotherapy with and without bevacizumab

DETAILED DESCRIPTION:
Subjects will be randomized in a 1:1 ratio to receive either Test Regimen or Comparator Regimen as the first-line treatment for advanced cervical cancer. Subjects will receive study therapy Q3W until progression of the disease or signs of unacceptable toxicity. In the absence of dose-limiting toxicity chemotherapy should be continued for at least 6 cycles, then, upon Investigator's decision and/or subjects' wish, the use of chemotherapy can be stopped while maintenance therapy with BCD-100/Placebo with or without bevacizumab (depending on initial therapy choice) continues until disease progression.

ELIGIBILITY:
Inclusion Criteria:

1. Signing an IRB/EC-approved informed consent
2. Females ≥ 18 years of age on day of signing informed consent
3. Histologically confirmed squamous carcinoma of the cervix
4. Progressing thru or recurrent disease treated for curative intent or primary metastatic cervical cancer stage FIGO IVB
5. Agreement to newly obtained core or excisional biopsy of a tumor lesion not previously irradiated for determination of PD-L1 status prior to randomization (using archival biopsy material is only acceptable in subjects in whom obtaining a new sample is contraindicated)
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
7. For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or to use a contraceptive method with a failure rate of < 1% per year from the moment of signing informed consent, during the treatment period and at least 6 months after administration of the last dose of study drug. A woman is considered to be of childbearing potential if she is postmenarcheal, has not reached a postmenopausal state (≥ 12 continuous months of amenorrhea with no identified cause other than menopause), and has not undergone surgical sterilization (removal of ovaries, fallopian tubes, and/or uterus). Examples of contraceptive methods with a failure rate of < 1% per year include but are not limited to bilateral tubal ligation and/or occlusion, male sterilization, and intrauterine devices. The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical study and the preferred and usual lifestyle of the subject. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) is not acceptable method of contraception.

Exclusion Criteria:

1. Indications for potentially curative treatment (surgery or radiation therapy)
2. Prior systemic treatment for recurrent, secondarily progressive or initially metastatic disease
3. Previous use of chemotherapy other than initial treatment for curative intent (e.g. chemotherapy used concurrently with radiation therapy, neoadjuvant or consolidation chemotherapy cycles before radiotherapy or 2 chemotherapy cycles after completion of chemoradiotherapy are allowed)
4. Contraindications to cisplatin, carboplatin, paclitaxel, or bevacizumab
5. Known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Participants with known brain metastases may participate provided that the brain metastases have been previously treated with radiotherapy or surgery only and are radiographically stable
6. Concomitant diseases or conditions which pose a risk of AE development during study treatment:

   1. uncontrolled hypertension, defined as systolic > 150 mm Hg or diastolic > 90 mm Hg;
   2. stable angina functional class III-IV;
   3. unstable angina or myocardial infarction less than 6 months prior to randomization;
   4. NYHA Grade III-IV congestive heart failure;
   5. serious cardiac arrhythmia requiring medication (subjects with asymptomatic atrial fibrillation can be enrolled if controlled ventricular rate);
   6. atopic asthma, Stage III-IV COPD, angioedema;
   7. severe respiratory failure;
   8. any other diseases which pose unacceptable risk of AE development during study treatment in Investigator's opinion.
7. Active or known or suspected autoimmune disease (subjects with Type 1 diabetes mellitus, hypothyroidism only requiring hormone replacement, or skin disorders (vitiligo, psoriasis, or alopecia) not requiring systemic treatment are permitted to enroll).
8. Condition requiring systemic treatment with either corticosteroids or other immunosuppressive medications within 14 days prior to randomization.
9. History of (non-infectious) pneumonitis that required corticosteroids or current pneumonitis
10. Neutrophils <1500/mcl or platelets <100 000/mcl or hemoglobin <90 g/l.
11. Creatinine ≥ 1.5 x UNL.
12. Bilirubin ≥ 1.5 x UNL (excluding Gilbert's syndrome if bilirubin < 50 µmol/l) or AST/ALT ≥ 3 x UNL (excluding subjects with liver metastases if AST/ALT < 5 x UNL) or alkaline phosphatase ≥ 2.5 x UNL.
13. Chemotherapy or radiation therapy less than 28 days prior to randomization.
14. Major surgery procedure less than 28 days prior to randomization.
15. Previous use of PD-1/PD-L1/PD-L2 agent or another agent directed to stimulatory or co-inhibitory T-cell receptor (e.g. CTLA-4, OX 40, CD137).
16. Previous use of VEGF/VEGFR inhibitors, including bevacizumab, ramucirumab, aflibercept and tyrosine kinase inhibitors.
17. Prior invasive malignancy with any evidence of disease within the last 3 years. Subjects with non-melanoma skin cancer or carcinoma in situ (e.g. breast cancer) who have undergone potentially curative therapy are not excluded.
18. Pre-existing clinically significant (≥ grade 2) peripheral neuropathy or hearing impairment
19. Any conditions or circumstances that limit subject's ability to comply with protocol requirements
20. Active hepatitis B, active hepatitis С or history of positive HIV.
21. Active infection requiring therapy or systemic antibiotics use less than 14 days prior to enrollment. Severe infections within 28 days prior to first study drug administration.
22. Administration of a live vaccine within 28 days prior to enrollment
23. Current using of another investigational device or drug study, or less than 30 days since ending of using of another investigational device or drug study
24. Life expectancy less than 12 weeks
25. Significant adverse events (AE) of previous therapy excluding chronic and/or irreversible events which cannot affect study drug safety evaluation (e.g. alopecia)
26. Known hypersensitivity or allergy to paclitaxel, cisplatin, carboplatin, bevacizumab, BCD-100 or any of their excipients. Known hypersensitivity or allergy to drugs derived from Chinese hamster (CHO) ovary cells or history of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins.
27. Pregnancy or breast-feeding

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 316 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | 3 years
  The time from the date of randomization until death

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) per RECIST 1.1 | 3 years
  The time from the date of randomization until progression of disease according to RECIST 1.1 criteria or death
Progression-Free Survival (PFS) per iRECIST | 3 years
  The time from the date of randomization until progression of disease according to iRECIS criteria or death
Overall Response Rate per (ORR) RECIST 1.1 | 1 year
  The percentage of the participants who have a Complete Response or a Partial Response as assessed by a blind independent central reviewer per RECIST 1.1
Overall Response Rate (ORR) per iRECIST | 1 year
  The percentage of the participants who have a Complete Response or a Partial Response as assessed by a blind independent central reviewer per iRECIST
Disease Control Rate (DCR) | 1 year
  The percentage of the participants who have a Complete Response, a Partial Response or a Stable DIsease as assessed by a blind independent central reviewer
Time to Response (TTR) | 1 year
  TTR will be calculated from the randomization date
Duration of Response (DOR) | 1 year
  DOR will be calculated from the moment of registration of response till event (progression or death)

CONTACTS AND LOCATIONS:
Overall Officials: Yulia N Linkova, MD, PhD, Study Director — Director of Clinical Development Department, BIOCAD
Locations (26):
- Shanghai Tenth People's Hospital, Shanghai, China
- Georgia (8):
  - High technology Hospital Medcenter, Batumi
  - Acad. F.Todua Medical center "Research institute of Clinical Medicine", Tbilisi
  - High Technology Medical Centre, University Clinic, Tbilisi
  - Institute for Personalized Medicine Ltd., Tbilisi
  - Institute of Clinical Oncology, Tbilisi
  - LEPL First University Clinic of Tbilisi State Medical University, Tbilisi
  - Multiprofile Clinic Consilium Medulla, Tbilisi
  - Neo Medi, Tbilisi
- Russia (16):
  - City Hospital No. 5, Barnaul
  - Krasnoyarsk Regional Clinical Oncological Dispensary named after A.I. Kryzhanovsky, Krasnoyarsk
  - Moscow Clinical Scientific and Practical Center named A.S. Loginova, Moscow
  - N.N. Blokhin National Medical Research Center of Oncology (2), Moscow
  - State Health Care Institution "Moscow City Oncology Hospital № 62" Moscow Health Department, Moscow
  - Murmansk Regional Clinical Hospital named after P.A. Bayandina, Murmansk
  - Clinical Oncology Dispensary, Omsk
  - LLC "New Clinic", Pyatigorsk
  - AV Medical Group, Saint Petersburg
  - JSC "Modern Medical Technologies", Saint Petersburg
  - N.N. Petrov National Medical Research Center of Oncology (2), Saint Petersburg
  - Saint-Petersburg Petersburg Clinical Scientific and Practical Center for Specialized Types of Medical Care (Oncological), Saint Petersburg
  - Federal State Educational Institution of Higher Professional Education "Mordovia State University N.P. Ogareva ", Saransk
  - Stavropol Regional Clinical Oncology Center, Stavropol
  - Regional Clinical Oncology Hospital, Yaroslavl
  - Sverdlovsk Regional Oncology Center, Yekaterinburg
- Memorial Şişli Istanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No